CLINICAL TRIAL: NCT04499001
Title: Effect of Pharmaceutical Consultations Just Before Rheumatology Consultations on Improving Knowledge and Skills for Patients With Inflammatory Arthritis Treated With Subcutaneous Biologic DMARDs
Brief Title: Effect of Pharmaceutical Consultations Just Before Rheumatology Consultations on Improving Knowledge and Skills for Patients With Inflammatory Arthritis With Subcutaneous Biologic DMARDs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Cécile Bottois, Principal Investigator, Hôpital Cochin
Other Study IDs: 2020-A01380-39
Record Dates: First submitted 2020-07-22; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Arthritis, Rheumatoid; Spondyloarthritis; Biological Therapy
Keywords: knowledge; safety skills; pharmaceutical consultation
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pharmacist's consultation — Information about bDMARDs management.

SUMMARY:
There is a lack of knowledge among patients concerning their treatment with bDMARDs. To increase knowledge and safety skills, patient education is essential.

The aim of this study is to assess the impact of a pharmacist's educational interview on on knowledge and safety skills to bDMARDs in patients with inflammatory arthritis.

DETAILED DESCRIPTION:
This is an observational, controlled, open-label and monocentric study. 60 patients are planned to be included.

Knowledge are assessed three time by self-administered questionnaire:

at baseline before the pharmacist's educational interview at three months apart at six months apart

One primary end-point is defined:

the changes from baseline to M3 and M6 in the patients' knowledge score about subcutaneous bDMARD management (self-administered questionnaire, Biosecure)

As secondary end-points, the changes from baseline to M3 and M6 in patients' adherence, patients' satisfaction regarding the pharmacists' intervention and the effect of the interview on rate of patients treated by biosimilar are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand and communicate in French and comply with the requirements of the study and must give his agreement (non-opposition) before any study assessment is performed.
* Patient at least 18 years of age
* Patient with inflammatory arthritis (rheumatoid arthritis or ankylosing spondylitis or other)
* Admission in medical consultation in the rheumatology department
* Patient treated with subcutaneous biologic DMARDs (Tocilizumab, Adalimumab, Etanercept, Golimumab, Certolizumab, Abatacept, Sarilumab, Ustekinumab, Ixekizumab, Anakinra)

Exclusion Criteria:

* Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from completing the study per protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with subcutaneous bDMARDs with inflammatory arthritis admitted in medical consultation in the rheumatology department
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in bDMARDS knowledge and skills at 3 and 6 months in patients who received a pharmaceutical consultation | 6 months of follow-up
  Knowledge level and score comparison (good or moderate or bad knowledge) evaluated by self-questionnaire (Biosecure) from baseline to M3 and M6 after the pharmaceutical consultation.
  Biosecure : Minimum = 0 ; Maximum = 100 Good knowledge > 84 Moderate knoledge : 64 to 84 Bad knowledge < 64
  Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change in bDMARDS adherence at 3 and 6 months in patients who received a pharmaceutical consultation | 6 months of follow-up
  Adherence level comparison (high or low adherence) evaluated by self-questionnaire, Compliance Questionnaire for Rheumatology (CQR-5) from baseline to M3 and M6 after the consultation.
  High adherence means a better outcome.
Satisfaction of patients on the pharmaceutical interview 3 months apart | 3 months of follow-up
  Assessment of patients' satisfaction on the pharmaceutical interview at 3 months of the consultation.
Change in rate of patients treated by biosimilar after the pharmaceutical consultation | 6 months of follow-up
  Comparison of patient treated by biosimilar rate from baseline to M3 and M6 after the consultation

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Bottois, Dr, Principal Investigator — Hôpital Cochin
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No